CLINICAL TRIAL: NCT02306746
Title: The Augmented Versus Routine Approach to Giving Energy Trial: A Randomised Controlled Trial
Brief Title: The Augmented Versus Routine Approach to Giving Energy Trial
Acronym: TARGET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZIC-RC/MC001
Record Dates: First submitted 2014-11-11; First posted 2014-12-03 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Critical Illness
Keywords: Enteral nutrition; randomised control trial; Critical care; Outcome
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TARGET protocol EN 1.5 kcal/mL (Experimental): Enteral (EN) feed 1.5 kcal/mL. The goal rate for administration of TARGET protocol EN is 1ml/kg/hr. To calculate the goal rate, weight is based on ideal body weight.
  Interventions: Dietary Supplement: TARGET protocol EN 1.5 kcal/mL
- TARGET protocol EN 1.0 kcal/mL (Active Comparator): Enteral feed 1.0 kcal/mL The goal rate for administration of TARGET protocol EN is 1ml/kg/hr. To calculate the goal rate, weight is based on ideal body weight.
  Interventions: Dietary Supplement: TARGET protocol EN 1.0 kcal/mL

INTERVENTIONS:
Dietary Supplement: TARGET protocol EN 1.5 kcal/mL — Enteral feed 1.5 kcal/mL
  Arms: TARGET protocol EN 1.5 kcal/mL
Dietary Supplement: TARGET protocol EN 1.0 kcal/mL — Enteral feed 1.0 kcal/mL
  Arms: TARGET protocol EN 1.0 kcal/mL

SUMMARY:
Nutrition therapy is an essential standard of care for all critically ill patients who are mechanically ventilated and remain in the intensive care unit for more than a few days.

The investigators plan to conduct a 4,000 patient, double-blind, randomised controlled trial to determine if augmentation of calorie delivery using energy dense enteral nutrition in mechanically ventilated patients improves 90 day survival when compared to routine care.

DETAILED DESCRIPTION:
Each year around 130,000 Australians are admitted to ICU at a daily cost of approximately $4000 per patient. Their care consumes close to 3 billion dollars per year. These critically ill patients are the sickest in the hospital. They require substantial resources and multiple interventions. Some die and many of those who survive have delayed and compromised functional recovery which can persist for months or years.

Nutrition therapy is an essential standard of care for all ICU patients who are mechanically ventilated and remain in ICU for more than a few days. Enteral nutrition (via a nasogastric tube) is usually initiated within 24 hours of ICU admission with a formula containing 1 kcal/ml and prescribed at an approximate rate of 1 ml/kg/hour. However, standard enteral nutrition practice typically results in the delivery of only ~60% of the full-recommended calorie requirement.

Although prescribed calories can reliably be delivered using the intravenous route, the enteral route is preferred for a number of reasons and is recommended by all nutrition guidelines as first-line therapy. In particular, enteral nutrition is more physiological, less costly and associated with fewer infective complications. Delivery of nutrient into the gut also has beneficial effects on subsequent gut function and may reduce ongoing sepsis which can be fuelled by the movement of gut flora through a permeable mucosa that has not been exposed to nutrient. Intravenous nutrition is accordingly, generally used only when enteral feeding is impossible, or persistently limited. Although supplementing enteral with intravenous nutrition can increase calorie delivery, this has not been shown to have a therapeutic benefit and may worsen important clinical outcomes. This may be because adverse effects associated with intravenous nutrition counteract the benefits of increased calorie delivery.

Previous trials support the concept that optimising nutrition in the critically ill will improve outcome, however, the evidence is limited, inclusive and generally of low quality. It is extraordinary that there is not better (Level I) evidence to inform nutrition management in critically ill patients given the frequency of the intervention, the biologic rationale, the high mortality following ICU admission, the frequency of muscle wasting and the poor functional outcomes in survivors. This is especially true given the low cost of enteral nutrition (~$23/day).

The investigators recently completed pilot study clearly achieved all the key criteria which, for a pharmaceutical product, would lead to a phase III trial, namely: 1. feasibility; 2. safety; 3. separation; 4. excellent recruitment rate; 5. successful blinding; 6. a signal for benefit.

A definitive study must now be done to establish whether 90-day survival and functional outcomes following critical illness may be improved by increased calorie delivery.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and receiving mechanical ventilation
* About to commence enteral nutrition or enteral nutrition commenced within the previous12 hours
* Expected to be receiving enteral nutrition in ICU until at least the day after tomorrow

Exclusion Criteria:

* Any Enteral Nutrition (EN) or Parenteral Nutrition (PN) received for >12 hours in this ICU admission
* Treating clinician considers the EN goal rate (i.e.1ml/kg of ideal body weight per hour) to be clinically contraindicated e.g. requirement for fluid restriction
* Requirement for specific nutritional therapy as determined by the treating doctor or dietitian i.e. TARGET protocol EN not considered to be in the best interest of the patient
* Death is deemed to be imminent or inevitable during this admission and either the attending physician, patient or substitute decision maker is not committed to active treatment
* The patient has an underlying disease that makes survival to 90 days unlikely
* ≥ 15% burns
* Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Day 90
  Mortality status

SECONDARY OUTCOMES:
Mortality | At hospital discharge an average of 28 days
  Mortality status
Mortality | Day 28
  Mortality status
Time from randomisation until death | Day 180
  Mortality status
Number of days alive and not in ICU | Day 28
  Mortality status
Number of days alive and not in hospital | Day 28
  Mortality status
Ventilator free days | Day 28
  Organ support status
Proportion of patients receiving vasopressor support | Day 28
  Organ support proportion
Vasopressor free days | Day 28
  Organ support status
Proportion of patients receiving any renal replacement therapy | Day 28
  Organ support proportion
Renal replacement therapy free days | Day 28
  Organ support status
Proportion of patients with positive blood cultures | Day 28
  Blood stream infection proportion
Proportion of patients requiring intravenous antimicrobials | Day 28
  Patients requiring intravenous antimicrobials
Mortality | Day 180
  Mortality status
Quality of life assessment | Day 180
  European Quality of Life 5 Dimensions
Functional outcomes for patients under 65 years in the work force | Day 180
  Questions from the Australian Labour Force Survey
Functional outcomes for patients under 65 years and not in the work force and patients 65 years and over living dependently | Day 180
  World Health Organization Disability Assessment Schedule 2.0
Functional outcomes for patients 65 years and over living independently | Day 180
  Adelaide Activities Profile
Cause-specific mortality | Day 90
  Mortality status

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Peake, MD, Study Chair — University of Adelaide
Locations (46):
- Australia (34):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Gosford Hospital, Gosford, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Royal North Shore Hosptial, Sydney, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Concord Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Logan Hospital, Brisbane, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Royal Adelaide Hosptial, Adelaide, South Australia
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Lyell McEwin, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Bendigo Hospital, Bendigo, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Frankston Hosptial, Frankston, Victoria
  - University Hosptial Geelong, Geelong, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Sunshine Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Monash Health Dandenong Hospital, Melbourne, Victoria
  - Bunbury Hospital, Bunbury, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - St John of God Hospital Murdoch, Perth, Western Australia
- New Zealand (12):
  - North Shore Hospital, Auckland
  - Auckland City Hospital Cardiovascular Intensive Care Unit, Auckland
  - Auckland City Hospital Department of Critical Care Medicine, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Hawkes Bay Fallen Soldiers Memorial Hospital, Hastings
  - Hutt Valley Hospital, Lower Hutt
  - Nelson Hospital, Nelson
  - Rotorua Hospital, Rotorua
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wittholz K, Fetterplace K, Chapple LA, Ridley EJ, Finnis M, Presneill J, Chapman M, Peake S, Bellomo R, Karahalios A, Deane AM. Six-month outcomes after traumatic brain injury in the Augmented versus Routine Approach to Giving Energy multicentre, double-blind, randomised controlled Trial (TARGET). Aust Crit Care. 2025 Mar;38(2):101116. doi: 10.1016/j.aucc.2024.09.001. Epub 2024 Oct 10. PMID 39389845
- [Derived] Arunachala Murthy T, Chapple LS, Lange K, Marathe CS, Horowitz M, Peake SL, Chapman MJ. Gastrointestinal dysfunction during enteral nutrition delivery in intensive care unit (ICU) patients: Risk factors, natural history, and clinical implications. A post-hoc analysis of The Augmented versus Routine approach to Giving Energy Trial (TARGET). Am J Clin Nutr. 2022 Aug 4;116(2):589-598. doi: 10.1093/ajcn/nqac113. PMID 35472097
- [Derived] TARGET Investigators, for the ANZICS Clinical Trials Group; Chapman M, Peake SL, Bellomo R, Davies A, Deane A, Horowitz M, Hurford S, Lange K, Little L, Mackle D, O'Connor S, Presneill J, Ridley E, Williams P, Young P. Energy-Dense versus Routine Enteral Nutrition in the Critically Ill. N Engl J Med. 2018 Nov 8;379(19):1823-1834. doi: 10.1056/NEJMoa1811687. Epub 2018 Oct 22. PMID 30346225
- See also: Statistical analysis plan publication, March 2018 — https://www.ncbi.nlm.nih.gov/pubmed/29458317
- See also: Protocol publication, March 2018 — https://www.ncbi.nlm.nih.gov/pubmed/29458316